CLINICAL TRIAL: NCT02283606
Title: Sonoelastography of the Uterine Cervix Before Induction of Labor
Acronym: SUCI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Rami Aviram, MD, Meir Medical Center
Other Study IDs: 0154-14-MMC
Record Dates: First submitted 2014-10-26; First posted 2014-11-05 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Accuvix SnonAce UGEO — vaginal ultrasonography

SUMMARY:
The investigators aim to measure sonoelastographically the elasticity of the uterine cervix in pregnant patients at term before induction of labor and compare between patients with successful and failed inductions.

DETAILED DESCRIPTION:
Softening of the uterine cervix in pregnant patients at term causes changes in its elasticity.these changes may affect success or failure in induction of labor.The elasticity of the uterine cervix is usually evaluated clinically and subjectively by vaginal examination (bishop's score) which is not very predictive.We aim to measure the elasticity quantitatively and objectively.The difference in strain, in the area of the internal os , is often illustrated by a color map, where low stiffness (soft tissue) is indicated in red, middle stiffness is in green and high stiffness (hard tissue) is in blue.The color maps will be compared between patients with successful and failed inductions.

ELIGIBILITY:
Inclusion Criteria:

* pregnant patients before induction of labor

Exclusion Criteria:

* pregnant patients undergoing caesaren section following induction of labor not in active labor

Ages: 20 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 20-44 years old pregnant patients
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Elasticity of the uterine cervix as measured sonoelastographically in successful and failed inductions of labor | 48-72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Rami Aviram, MD, Principal Investigator — Meir Medical Center